CLINICAL TRIAL: NCT03253445
Title: Individual, Acceptance and Commitment Therapy (ACT) in Smoking Cessation for People With Schizophrenia: a Randomized Controlled Trial
Brief Title: Individual Acceptance and Commitment Therapy (ACT) for Smoking Cessation for Schizophrenic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Yim Wah Mak, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ACTSP01032016
Record Dates: First submitted 2016-03-18; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; acceptance and commitment therapy; ACT; schizophrenic patients; hostel setting; randomised controlled trial
MeSH Terms: conditions — Smoking Cessation | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acceptance and commitment therapy (Experimental): All participants are given a brief educational talk on encouraging quitting smoking, a self-help leaflet on smoking cessation and an additional 10-session face-to-face ACT on a weekly basis.
  Interventions: Behavioral: Acceptance and commitment therapy
- Control (Placebo Comparator): All participants are given a brief educational talk on encouraging quitting smoking , a self-help leaflet on smoking cessation and 10-sessions of face-to-face social support on a weekly basis.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — All participants are given a brief educational talk on encouraging quitting smoking (about 5 mins) and a self-help leaflet on smoking cessation. Ten sessions of face-to-face ACT individually will additionally be provided by trained therapists on a weekly basis. Each session will last about 20-30 minutes. The therapy is guided by ACT smoking cessation protocols based on relevant literature (Gifford et al 2004, 2011; Bricker, 2010).
  Other Names: ACT
  Arms: Acceptance and commitment therapy
Other: Control — All participants are given a brief educational talk on encouraging quitting smoking (about 5 mins) and a self-help leaflet on smoking cessation. Ten sessions of face-to-face Social Support will additionally be provided on a weekly basis. Each session will last about 5 minutes.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the efficacy of using Acceptance and commitment therapy for smoking cessation for schizophrenic patients.

DETAILED DESCRIPTION:
Background: Amongst people with mental disorders, the prevalence of smoking has been reported to be the highest among people with schizophrenia, ranging from 54%-90%. It is more than two to three times (20%-30%) of the general population. The co-occurrence of schizophrenia and smoking will lead to a higher chance of smoking-related diseases such as cardiovascular disease, liver diseases and reduced life expectancy. Currently, there is a large gap in knowledge regarding smoking cessation in people with schizophrenia; there has been few studies examining non-pharmacological interventions in smoking cessation on people with schizophrenia. Acceptance and commitment therapy (ACT) for mental health disorders has found that it has in general positive outcomes for the clients; improvements were consistently found in a number of studies. ACT is more encouraging compared to traditional methods of smoking cessation, where the individual is seen to be at fault for the habit. To date, no randomized trial has been conducted to compare the effects of ACT in smoking cessation among people with schizophrenia.

Objective: To evaluate the efficacy of Acceptance and Commitment Therapy (ACT) in enhancing smoking cessation among people with schizophrenia living in the community.

Design: This is a randomised controlled trial. Individual, face to face, assessor-blinded with assessments will be conducted before intervention, after intervention, and at the 6th and 12th month after the initial session of ACT intervention.

Participants and setting: 160 individuals aged 18 years or older, currently smoking but not undergoing any smoking cessation or similar programme, who were diagnosed with schizophrenia and were referred to 4 community-based mental health rehabilitation settings by medical doctors will be included in this trial.

Using the Six Core Processes in Intervention (Flaxman, Blackledge & Bond, 2010) Acceptance By acceptance, ACT does not mean by the traditional sense of "letting go", "admitting faith passively", or "do something after acknowledging the facts". Since psychological avoidance toward distress, which can be unfavorable thoughts, emotions, will inevitably push individual to evade such experiences, ACT attacks the problem by accepting the psychological distress as it is, without distorting, interpreting or re-interpreting it through verbal constructs.

Defusion Patients frequently, if not inevitably, fall into the trap of fusing their thoughts and appraisals with their self-concept. They are often so identified with the internal dialogues that whenever a thought of judging themselves arise, they treat them as a valid statement of evaluation on themselves. Cognitive defusion aims at creating a space between the thought and its relation with the individual, with the effect that the words, thoughts, and emotions are down-valued as a reference rather than a valid description of who we are.

Self as context Our sense of self is often derived from our experienced thoughts, emotions, memories and physical sensations. This is called the self-as-content and is a readily accessible self-concept most of us would refer to. By addressing the above experience, especially the more frequent ones, we draw the conclusion that we are the person defined by them. On the contrary, ACT adopts the notion of self-as-context and defines the self as that stable, ever-present part of you that notices the transient thoughts, emotions, memories and sensations that enter in and out of awareness. When the self-as-context is embraced, the self is no longer defined as the various thoughts, feelings, and sensations, but as the person who is having or noticing those experiences. Although ACT makes no attempt to discern which one is a better representation of the self, it does appreciate self-as-context as a way to examine the distance between those internal experiences and the self.

Contact with the Present Moment Making a closer contact with the present moment is the key to seeing how effectively or ineffectively what we are behaving in the moment, and that places us in a better position to change our behaviors as well as a higher motivation to do so. However, thoughts are always pulling us away from the present moment and we are either in the past or future. In fact, thoughts are about anything and everything except now.

Values Values are perhaps the most powerful reinforcers in driving us to our goal and at the same time a valuable asset for individuals who are trying to live what they expect from life. Instead of swamping oneself in numerous problems, issues, regrets, and longings, values provide a powerful drive for patients to act according to what they want to become. Therapist, on the other hand, have a consistent measure as to the way the patients have to live up to their own expectations. Still more, therapist and patients are to endeavor collaboratively in working out the qualities in realizing patients' values.

Committed Action If value is the train, commitment is the fuel that drives the person forward. Value, together with commitment, is a non-binding guideline that points to the way an individual can act. Therapist, on the other hand, is supposed to reinforce and encourage behaviors that are consistent with the values. Any behaviors inconsistent with the values are to be accepted as they are in a non-judgmental attitude, and the patient is encouraged to choose again in accordance to his values. Commitment is not only viewed as a promise but also actions that realize what one believes and upholds.

Competency of therapist:

The following are extracted from the core competencies self rating form posted at the website of Association for Contextual Behavioral Science (Luoma, n.d.).

Basic competency in ACT The therapist is able to take heed of the patient's schizophrenic background and introduce the concepts and skills of ACT in a simple language that is compatible with the level of cognition and intelligence of the patient.

The therapist helps the patient to realize his beliefs, thoughts, desires, fears and worries with smoking cessation.

The therapist assists the patient in addressing in-depth his/her motivations and values regarding smoking cessation.

The therapist is capable of leading the patient to apprehend the futility of the attempts to control the cravings and accept the urges as it is without necessarily yielding to them.

By guiding the patient to see the hopelessness of controlling craving, the therapist is able to guide the patient to the ultimate solution-doing nothing, i.e., the mindfulness strategy of observing the cravings without the need to do anything.

The therapist assists the patient to bring about actions in executing his/her values in a practical manner amidst even the most unfavorable circumstances as perceived by the patient.

The therapist is able to master the six core processes of ACT and uses them flexibly by the flow of the therapy and the need of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or above;
2. diagnosed with schizophrenia;
3. referred by medical doctors;
4. currently smoking, i.e. have at least one cigarette per day in the past month,
5. willing to take part in a face-to-face individual intervention program in changing smoking behaviors such as smoking cessation, reduction of cigarette consumed, or the relief of withdrawal symptoms.
6. able to communicate in Cantonese.

Exclusion Criteria:

1. disorientation, developmental disabilities, and/or organic conditions that will inhibit his/her understanding and participation in the therapeutic process,
2. diagnosis of alcohol or drug dependence in the preceding year of recruitment or,
3. medication regime revised in the last 3 months or,
4. current participation in another smoking cessation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Self-report of not having smoked for the past 7 days | At 6th month after the initial intervention
  Self-report of not having smoked for the past 7 days at 6th month after initial intervention

SECONDARY OUTCOMES:
Self-report of not having smoked for the past 7 days | At 12th month after the initial intervention
  Self-report of not having smoked for the past 7 days at 12th month after initial intervention
Self-report of not having smoked for 7 days at 6th month after initial intervention, as validated by exhaled carbon monoxide test | At 6th month after the initial intervention
  Using exhaled carbon monoxide test to validate self-report of not having smoked for 7 days at 6th month after initial intervention
Self-report of not having smoked for 7 days at 6th month after initial intervention, as validated by urinary cotinine test | At 6th month after the initial intervention
  Using urinary cotinine test to validate self-report of not having smoked for 7 days at 6th month after initial intervention
Self-report of not having smoked for 7 days at 12th month after initial intervention, as validated by urinary cotinine test | At 12th month after the initial intervention
  Using urinary cotinine test to validate self-report of not having smoked for 7 days at 12th month after initial intervention
Forward progression on stages of readiness in smoking cessation | At 6th month after the initial intervention
  Self-report of forward progression on stages of readiness in smoking cessation. Prochaska's Transtheoretical Model of behavior change is used to assess the stages of readiness in smoking cessation
Increasing psychological flexibility | At 6th month and 12th month after the initial intervention
  Acceptance and Action Questionnaire - II (AAQ-II) is used to assess the psychological flexibility of the participants

CONTACTS AND LOCATIONS:
Overall Officials: YW Mak, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University; AY Loke, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Twohig MP, Crosby JM. Acceptance and commitment therapy as a treatment for problematic internet pornography viewing. Behav Ther. 2010 Sep;41(3):285-95. doi: 10.1016/j.beth.2009.06.002. Epub 2010 Jan 28. PMID 20569778
- [Background] Flaxman PE, Blackledge JT, Bond FW. Acceptance and commitment therapy: Distinctive features. London & New York: Routledge; 2002.
- [Background] Bricker JB, Mann SL, Marek PM, Liu J, Peterson AV. Telephone-delivered Acceptance and Commitment Therapy for adult smoking cessation: a feasibility study. Nicotine Tob Res. 2010 Apr;12(4):454-8. doi: 10.1093/ntr/ntq002. Epub 2010 Feb 8. PMID 20142417
- [Background] Gifford EV, Kohlenberg BS, Hayes SC, Pierson HM, Piasecki MP, Antonuccio DO, Palm KM. Does acceptance and relationship focused behavior therapy contribute to bupropion outcomes? A randomized controlled trial of functional analytic psychotherapy and acceptance and commitment therapy for smoking cessation. Behav Ther. 2011 Dec;42(4):700-15. doi: 10.1016/j.beth.2011.03.002. Epub 2011 May 25. PMID 22035998
- [Background] Gifford EV, Kohlenberg BS, Hayes SC, Antonuccio DO, Piasecki MM, Rasmussen-Hall ML, et al. Acceptance based treatment for smoking cessation. Behav Ther. 2004;35(4):689-705. doi: 10.1016/S0005-7894(04)80015-7. Epub 2006 Mar 3.
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700